CLINICAL TRIAL: NCT05296915
Title: Bulimia Nervosa e Binge Eating Disorder: Strategie Terapeutiche a Confronto
Brief Title: Bulimia Nervosa and Binge Eating Disorder: Comparing Therapeutic Strategies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DIGEST
Record Dates: First submitted 2022-03-16; First posted 2022-03-25 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-03

CONDITIONS: Bulimia Nervosa; Binge-Eating Disorder
Keywords: Bulimia Nervosa; Eating disorders; rTMS; CBT-E; tVNS; EEG
MeSH Terms: conditions — Bulimia Nervosa; Binge-Eating Disorder; Feeding and Eating Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: In order to achieve the objectives of the research project, we will perform a national, monocentric interventional on a medical device study, controlled in 3 parallel and randomized groups with a 1:1:1 allocation ratio.
Who Masked: Investigator
Masking Description: Personnel responsible for HRV analysis and determination of inflammatory biomarker levels will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tVNS + CBT-E group (Experimental): N=10 Interventional group with transcutaneous stimulation of the auricular branch of the vagus nerve associated with targeted cognitive-behavioral therapy (following the CBT-E protocol, CG Fairburn - 2010.
  Interventions: Device: tVNS; Behavioral: CBT-E
- rTMS + CBT-E group (Experimental): N=10 Interventional group with repetitive transcranial magnetic stimulation associated with targeted cognitive-behavioral therapy (following the CBT-E protocol, CG Fairburn - 2010.).
  Interventions: Device: rTMS; Behavioral: CBT-E
- Only CBT-E group (Experimental): N=10 Group with only cognitive-behavioral therapy of eating disorders.
  Interventions: Behavioral: CBT-E

INTERVENTIONS:
Device: tVNS — An electric current with a frequency of 25 Hz (Figure 2) will be applied to the cymba conca of the left ear through a specific device (VITOS, Cerbomed, Germany; CE marking). The stimulation intensity will be customized between 0.1 and 5 mA according to the sensitivity threshold of each participant. Patients will be instructed to perform tVNS at home for 4 non-consecutive hours per day for 12 weeks, in accordance with the protocol reported in the literature for the treatment of major depression.
  Other Names: Transcutaneous stimulation of the auricular branch of the vagus nerve associated
  Arms: tVNS + CBT-E group
Device: rTMS — The stimulation will be carried out with a TMS STM9000 system (Ates, Medica Device s.r.l., Italy) equipped with a 70 mm "butterfly" cooled coil. The stimulation protocol followed will be the one approved by the FDA for major depression, that is, a stimulation at the level of the left dorsolateral prefrontal cortex at an intensity equal to 120% of the motor threshold, at the frequency of 10hz. Each stimulation session will last 37.5 minutes, and will consist of 75 trains lasting 4 seconds, with a 26-second break between each train. During each session, a total of 3000 stimuli will be administered. The sessions will take place 5 days a week, from Monday to Friday, for 4 weeks, and for a total of 20 sessions of stimulation.
  Other Names: Repetitive transcranial magnetic stimulation
  Arms: rTMS + CBT-E group
Behavioral: CBT-E — Targeted cognitive-behavioral therapy following the CBT-E protocol (CG Fairburn - 2010. La terapia cognitivo-comportamentale dei disturbi dell'alimentazione. Firenze, Eclipsi; 2010.)
  Other Names: Cognitive-behavioral therapy - enanched

SUMMARY:
This study aims to assess the effectiveness of new neurostimulation techniques in patients with eating disorders.

The primary aim of our proposal is to test a reduction in symptoms of alteration of eating behaviors, such as always thinking about food or binge eating, in a sample of 30 patients, aged between 18 and 65, with diagnosis of Bulimia Nervosa or Binge Eating Disorder. Of these patients, 10 will undergo to a protocol of vagal transcutaneous stimulation in the ear (tVNS) and targeted cognitive-behavioral therapy (CBT-E), another 10 to a protocol of transcranial magnetic stimulation (rtms) and CBT-E and another 10 to a protocol of only tergeted CBT-E, comparing the results obtained in the three groups under study. Secondary purposes of this project are the assessment of the effects of auricular vagal transcutaneous stimulation and of transcranial magnetic stimulation on depressive symptoms associated with eating disorder, on the inflammatory profile, on cardiovascular autonomic control, neuronal excitability, functional connectivity and on the quality of life of these patients.

In order to achieve the objectives of this research project, we will perform a national, interventional on a medical device, monocentric study, controlled in 3 parallel and randomized groups with a 1:1:1 allocation ratio. 30 patients will be recruited at the Day Hospital of the Psychiatry Unit of the Fondazione.

DETAILED DESCRIPTION:
This study aims to assess the effectiveness of new neurostimulation techniques in patients with eating disorders.

To date, the management of these disorders is still difficult and few treatments have proven their effectiveness. According to most guidelines, management is typically multidisciplinary. The best validated and most frequently used treatment is the cognitive behavioral therapy enanched (CBT-E), a highly individualized psychological treatment designed to treat all diagnostic categories of eating disorders, addressing the common cognitive-behavioural mechanisms of maintaining shared and evolving psychopathology of eating disorders.

For Bulimia Nervosa (BN) and Binge Eating Disorder (BED), the serotoninergic antidepressants are the most frequently used pharmacological option (considering the frequent recurrence of depressive symptoms in comorbidity in the clinical population with eating disorders), which may improve symptoms in the medium term, but not allow complete remission. In this context, the development of alternative therapeutic strategies is crucial. Recently, several studies have described the important contribution of neurostimulation techniques (such as repetitive transcranial magnetic stimulation (rTMS), and vagal nerve stimulation (VNS)). Following the proven effectiveness, both rTMS and VNS have received official approval for the treatment of depression in Europe and United States. Neuroimaging studies have revealed that both of these neurostimulation techniques modulate the frontal-vagal network, the one with a top-down mechanism (rTMS) and the other with a bottom-up mechanism (VNS).

The neuromodulation influencing the functioning of the central nervous system (CNS) and the emotional/alimentary behavior, would offer an alternative (or complementary) intervention to psychotropic drugs and different psychological and nutritional approaches. Studies in the literature, conducted on patients with BN and BED, showed a significant improvement in symptomatology, in terms of "binge eating", after rTMS stimulation of the left dorsolateral prefrontal cortex (DLPFC). Instead, the effectiveness of vagal stimulation in the treatment of ED lies in the fact that the vagus nerve plays a fundamental role in mood and appetite regulation. Human studies report how tVNS stimulation produces a reduction in the effect of food cravings. Moreover, currently, in patients with ED, the determined effects of vagal non-invasive neurostimulation have not been compared with the effects of repetitive transcranial magnetic stimulation.

Therefore, the primary aim of our proposal is to test a reduction in symptoms of alteration of eating behaviors, such as always thinking about food or binge eating, in a sample of 30 patients, aged between 18 and 65, with diagnosis of Bulimia Nervosa or Binge Eating Disorder, according to the diagnostic criteria of DSM-V, and with a psychopathological framework of depression in comorbidity (cut-off ≥ 8 of the Hamilton Depression Rating Scale, HAM-D). Of these patients, 10 will undergo to a protocol of vagal transcutaneous stimulation in the ear (tVNS) and targeted cognitive-behavioral therapy (CBT-E), another 10 to a protocol of transcranial magnetic stimulation (rtms) and targeted cognitive-behavioral therapy (CBT-E) and another 10 to a protocol of only tergeted cognitive-behavioral therapy (CBT-E), comparing the results obtained in the three groups under study. Secondary purposes of this project are the assessment of the effects of auricular vagal transcutaneous stimulation and of transcranial magnetic stimulation on depressive symptoms associated with eating disorder, on the inflammatory profile, on cardiovascular autonomic control, neuronal excitability, functional connectivity and on the quality of life of these patients.

In order to achieve the objectives of this research project, we will perform a national, interventional on a medical device, monocentric study, controlled in 3 parallel and randomized groups with a 1:1:1 allocation ratio. 30 patients will be recruited at the Day Hospital of the Psychiatry Unit of the Fondazione.

Patients will be assigned by randomization to 3 different groups/treatments:

* tVNS+CBT-E group: 10 patients will be instructed to perform tVNS at home for 4 non-consecutive hours per day for 12 weeks with the tVNS VITOS device (already used in the Fondazione for the study tVNS2019 approved by the Milan Area 2 Ethics Committee on 19.02.2019 and with code 158_2019bis);
* rTMS+CBT-E group: 10 patients will participate in a total of 20 rTMS sessions lasting 40 minutes (5 sessions per week for 4 weeks) that will take place at the Day Hospital of the Psychiatry Unit of the Fondazione;
* CBT-E only group: 10 patients will proceed with only targeted cognitive behavioral therapy (CBT-E), following the CBT-E protocol CG Fairburn - 2010.

During the screening visit, provided by normal clinical practice, the inclusion and exclusion criteria and the diagnosis of Bulimia Nervosa and Binge Eating Disorder will be verified through a structured clinical interview planned for DSM-5 and personality disorders (by administration of the SCID-5 CV and PD scales by the physician). All patients will then be evaluated during 5 extra standard care visits. At each visit dietary behavior and any depressive symptoms will be evaluated through scales validated in Italian (Eating Disorder Examination, Eating Disorder Inventory, Eating Disorder Examination Questionnaire, Hamilton Depression Rating Scale and Beck Depression Inventory); cardiovascular variables will be recorded during clinostatism and orthostatism; a resting EEG and a during acute administration of transcranial magnetic stimulation EEG (TMS-EEG) will be recorded; participants will be asked to self-compile 2 questionnaires on the quality of life linked to health; finally a blood sample will be taken for the analysis of the inflammatory profile. For each patientd an Holter-ECG will be recorded lasting 72h following each visit. All the devices used in the study have already been purchased with university funds and have been taken over, labelled and coded by the Clinical Engineering of the Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico di Milano.

ELIGIBILITY:
Inclusion Criteria: patients diagnosed with Bulimia Nervosa or Binge Eating Disorder, according to the diagnostic criteria of DSM-V, with a psychopathological framework of depression in comorbidity (cut-off ≥ 8 of the Hamilton Depression Rating Scale, HAM-D), aged between 18 and 65 years.

Exclusion Criteria:

* Previous TMS sessions with significant side effects;
* Conditions leading to an increased risk of epilepsy or side effects in the context of transcranial magnetic stimulation (including personal or family history of epilepsy, cerebral ischemic events, neurological pathologies, neurosurgical interventions, orthopedic or vascular interventions in the head-neck district, major head trauma, migraine or severe headache);
* Presence of pacemakers, defibrillators, infusion pumps, neurostimulation implants (DBS, VNS), endovascular implants in the head-neck district, cochlear implants, cerebrospinal shunts, metal implants in the head-neck area ;
* Exposure to penetration of metal chips in the head-neck area;
* Presence of non-removable metal in the head-neck area (including tattoos, permanent make-up, piercing, excluding dental implants);
* Unstable sinus rhythm at ECG (Pace-Maker rhythm, atrial fibrillation, supra-/ventricular extrasystole);
* Chronic intake of β-blocker;
* Heart, respiratory, renal or hepatic failure and immunosuppression;
* Current hospitalization;
* State of pregnancy or lactation;
* Vestibular or balance problems;
* Positive personal history of schizophrenia or schizoaffective disorder;
* Substance or alcohol abuse in the last 6 months;
* Positive personal history of intellectual disability ("mental retardation");
* Refusal of informed consent by the patient.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Changing in dietary behaviour in terms of changes in Eating Disorder Examination scale score at T3 | 6 months from the start of treatment
  Effectiveness in changing dietary behaviour in terms of the EDE (Eating Disorder Examination) score difference between groups at T3. Great differences mean better clinical outcome.

SECONDARY OUTCOMES:
Incidence of acute effects of treatments in terms of difference between pre- and post-treatment | After 4 weeks of stimulation (T1)
  Incidence of acute effects of treatment with tVNS+CBT-E, rTMS+CBT-E or only CBT-E in patients with Eating Disorders in terms of difference between pre- and post-treatment for:
  * Variations in EDE-Q (Eating Disorder Examination Questionnaire) validated questionnaire scores.
  * Depressive symptoms: change in HAM-D and BDI-II scores.
  * Change in the systemic inflammatory profile: values of inflammatory serum proteins (IL-6, IL-1β, IL-4, IL-10, TNF-α and PCR) and microvesicles.
  * Changes in cardiovascular autonomic control: spectral power (ms2) and percentage (normalized units), over 250 beats, of the following frequency classes: very low frequency (VLF), low frequency (LF, 0.04-0.15 Hz) and high frequency (HF, 0.15-0.40 Hz). Percentage on 250 beats, of pattern 0V, 2LV and 2UV (symbolic analysis).
  * For TMS+EEG: variation of neuronal excitability patterns and functional connectivity and changes in quality of life in terms of total score of the CIA 3.0, PSQI validated questionnaires.
Incidence of acute effects of treatments in terms of difference between pre- and post-treatment | After 12 weeks of stimulation (T2)
  Incidence of acute effects of treatment with tVNS+CBT-E, rTMS+CBT-E or only CBT-E in patients with Eating Disorders in terms of difference between pre- and post-treatment for:
  * Variations in EDE-Q (Eating Disorder Examination Questionnaire) validated questionnaire scores.
  * Depressive symptoms: change in HAM-D and BDI-II scores.
  * Change in the systemic inflammatory profile: values of inflammatory serum proteins (IL-6, IL-1β, IL-4, IL-10, TNF-α and PCR) and microvesicles.
  * Changes in cardiovascular autonomic control: spectral power (ms2) and percentage (normalized units), over 250 beats, of the following frequency classes: very low frequency (VLF), low frequency (LF, 0.04-0.15 Hz) and high frequency (HF, 0.15-0.40 Hz). Percentage on 250 beats, of pattern 0V, 2LV and 2UV (symbolic analysis).
  * For TMS+EEG: variation of neuronal excitability patterns and functional connectivity and changes in quality of life in terms of total score of the CIA 3.0, PSQI validated questionnaires.
Incidence of long-term effects in terms of relapses and difference between T0 and T4. | After 12 months (T4) from enrollment
  Incidence of long-term effects of the three treatments (tVNS + CBT-E, rtms + CBT-E and CBT-E) in patients with BN and BED in terms of relapses and difference between T0 and T4 for the following indices:
  * Dietary behaviour: change in EDE and EDE-Q scores.
  * Depressive symptoms: change in HAM-D and BDI-II scores
  * Change in the systemic inflammatory profile: values of inflammatory serum proteins (IL-6, IL-1β, IL-4, IL-10, TNF-α and PCR) and microvesicles.
  * Changes in cardiovascular autonomic control: spectral power (ms2) and percentage (normalized units), over 250 beats, of the following three frequency classes: very low frequency (VLF), low frequency (LF, 0.04-0.15 Hz) and high frequency (HF, 0.15-0.40 Hz). Percentage on 250 beats, of pattern 0V, 2LV and 2UV (symbolic analysis).
  * TMS + EEG: Variation of neuronal excitability patterns and functional connectivity.
  * Changes in quality of life: total score of PSQI and CIA 3.0 validated questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Brambilla, Professor, Study Chair — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zabala MJ, Macdonald P, Treasure J. Appraisal of caregiving burden, expressed emotion and psychological distress in families of people with eating disorders: a systematic review. Eur Eat Disord Rev. 2009 Sep-Oct;17(5):338-49. doi: 10.1002/erv.925. PMID 19367608
- [Background] Treasure J, Duarte TA, Schmidt U. Eating disorders. Lancet. 2020 Mar 14;395(10227):899-911. doi: 10.1016/S0140-6736(20)30059-3. PMID 32171414
- [Background] Fairburn CG, Cooper Z, Doll HA, O'Connor ME, Bohn K, Hawker DM, Wales JA, Palmer RL. Transdiagnostic cognitive-behavioral therapy for patients with eating disorders: a two-site trial with 60-week follow-up. Am J Psychiatry. 2009 Mar;166(3):311-9. doi: 10.1176/appi.ajp.2008.08040608. Epub 2008 Dec 15. PMID 19074978
- [Background] Fairburn CG, Cooper Z, Doll HA, O'Connor ME, Palmer RL, Dalle Grave R. Enhanced cognitive behaviour therapy for adults with anorexia nervosa: a UK-Italy study. Behav Res Ther. 2013 Jan;51(1):R2-8. doi: 10.1016/j.brat.2012.09.010. Epub 2012 Oct 22. PMID 23084515
- [Background] Poulsen S, Lunn S, Daniel SI, Folke S, Mathiesen BB, Katznelson H, Fairburn CG. A randomized controlled trial of psychoanalytic psychotherapy or cognitive-behavioral therapy for bulimia nervosa. Am J Psychiatry. 2014 Jan;171(1):109-16. doi: 10.1176/appi.ajp.2013.12121511. PMID 24275909
- [Background] Dalle Grave R, Calugi S, Doll HA, Fairburn CG. Enhanced cognitive behaviour therapy for adolescents with anorexia nervosa: an alternative to family therapy? Behav Res Ther. 2013 Jan;51(1):R9-R12. doi: 10.1016/j.brat.2012.09.008. Epub 2012 Oct 4. PMID 23123081
- [Background] Dalle Grave R, Calugi S, Conti M, Doll H, Fairburn CG. Inpatient cognitive behaviour therapy for anorexia nervosa: a randomized controlled trial. Psychother Psychosom. 2013;82(6):390-8. doi: 10.1159/000350058. Epub 2013 Sep 20. PMID 24060628
- [Background] Dalle Grave R, Calugi S, El Ghoch M, Conti M, Fairburn CG. Inpatient cognitive behavior therapy for adolescents with anorexia nervosa: immediate and longer-term effects. Front Psychiatry. 2014 Feb 12;5:14. doi: 10.3389/fpsyt.2014.00014. eCollection 2014. PMID 24575055
- [Background] Tobaldini E, Carandina A, Toschi-Dias E, Erba L, Furlan L, Sgoifo A, Montano N. Depression and cardiovascular autonomic control: a matter of vagus and sex paradox. Neurosci Biobehav Rev. 2020 Sep;116:154-161. doi: 10.1016/j.neubiorev.2020.06.029. Epub 2020 Jun 26. PMID 32598983
- [Background] Iseger TA, van Bueren NER, Kenemans JL, Gevirtz R, Arns M. A frontal-vagal network theory for Major Depressive Disorder: Implications for optimizing neuromodulation techniques. Brain Stimul. 2020 Jan-Feb;13(1):1-9. doi: 10.1016/j.brs.2019.10.006. Epub 2019 Oct 10. PMID 31668983
- [Background] Thayer JF, Lane RD. Claude Bernard and the heart-brain connection: further elaboration of a model of neurovisceral integration. Neurosci Biobehav Rev. 2009 Feb;33(2):81-8. doi: 10.1016/j.neubiorev.2008.08.004. Epub 2008 Aug 13. PMID 18771686
- [Background] Van den Eynde F, Guillaume S. Neuromodulation techniques and eating disorders. Int J Eat Disord. 2013 Jul;46(5):447-50. doi: 10.1002/eat.22100. No abstract available. PMID 23658089
- [Background] Duriez P, Bou Khalil R, Chamoun Y, Maatoug R, Strumila R, Seneque M, Gorwood P, Courtet P, Guillaume S. Brain Stimulation in Eating Disorders: State of the Art and Future Perspectives. J Clin Med. 2020 Jul 23;9(8):2358. doi: 10.3390/jcm9082358. PMID 32717984
- [Background] Bodenlos JS, Kose S, Borckardt JJ, Nahas Z, Shaw, O'Neil PM, Pagoto SL, George MS. Vagus nerve stimulation and emotional responses to food among depressed patients. J Diabetes Sci Technol. 2007 Sep;1(5):771-9. doi: 10.1177/193229680700100524. PMID 19885147
- [Background] Calugi S, Sartirana M, Milanese C, El Ghoch M, Riolfi F, Dalle Grave R. The clinical impairment assessment questionnaire: validation in Italian patients with eating disorders. Eat Weight Disord. 2018 Oct;23(5):685-694. doi: 10.1007/s40519-018-0477-2. Epub 2018 Jan 24. PMID 29368290
- [Background] Curcio G, Tempesta D, Scarlata S, Marzano C, Moroni F, Rossini PM, Ferrara M, De Gennaro L. Validity of the Italian version of the Pittsburgh Sleep Quality Index (PSQI). Neurol Sci. 2013 Apr;34(4):511-9. doi: 10.1007/s10072-012-1085-y. Epub 2012 Apr 13. PMID 22526760
- [Background] Val-Laillet D, Aarts E, Weber B, Ferrari M, Quaresima V, Stoeckel LE, Alonso-Alonso M, Audette M, Malbert CH, Stice E. Neuroimaging and neuromodulation approaches to study eating behavior and prevent and treat eating disorders and obesity. Neuroimage Clin. 2015 Mar 24;8:1-31. doi: 10.1016/j.nicl.2015.03.016. eCollection 2015. PMID 26110109
- [Background] Steenbergen L, Sellaro R, Stock AK, Verkuil B, Beste C, Colzato LS. RETRACTED: Transcutaneous vagus nerve stimulation (tVNS) enhances response selection during action cascading processes. Eur Neuropsychopharmacol. 2015 Jun;25(6):773-8. doi: 10.1016/j.euroneuro.2015.03.015. Epub 2015 Mar 30. PMID 25869158
- [Background] De Risio L, Borgi M, Pettorruso M, Miuli A, Ottomana AM, Sociali A, Martinotti G, Nicolo G, Macri S, di Giannantonio M, Zoratto F. Recovering from depression with repetitive transcranial magnetic stimulation (rTMS): a systematic review and meta-analysis of preclinical studies. Transl Psychiatry. 2020 Nov 10;10(1):393. doi: 10.1038/s41398-020-01055-2. PMID 33173042
- [Background] Miller AH, Raison CL. The role of inflammation in depression: from evolutionary imperative to modern treatment target. Nat Rev Immunol. 2016 Jan;16(1):22-34. doi: 10.1038/nri.2015.5. PMID 26711676
- [Background] Kohler CA, Freitas TH, Maes M, de Andrade NQ, Liu CS, Fernandes BS, Stubbs B, Solmi M, Veronese N, Herrmann N, Raison CL, Miller BJ, Lanctot KL, Carvalho AF. Peripheral cytokine and chemokine alterations in depression: a meta-analysis of 82 studies. Acta Psychiatr Scand. 2017 May;135(5):373-387. doi: 10.1111/acps.12698. Epub 2017 Jan 25. PMID 28122130
- [Background] Arteaga-Henriquez G, Simon MS, Burger B, Weidinger E, Wijkhuijs A, Arolt V, Birkenhager TK, Musil R, Muller N, Drexhage HA. Low-Grade Inflammation as a Predictor of Antidepressant and Anti-Inflammatory Therapy Response in MDD Patients: A Systematic Review of the Literature in Combination With an Analysis of Experimental Data Collected in the EU-MOODINFLAME Consortium. Front Psychiatry. 2019 Jul 9;10:458. doi: 10.3389/fpsyt.2019.00458. eCollection 2019. PMID 31354538
- [Background] Reardon C, Murray K, Lomax AE. Neuroimmune Communication in Health and Disease. Physiol Rev. 2018 Oct 1;98(4):2287-2316. doi: 10.1152/physrev.00035.2017. PMID 30109819
- [Background] Borovikova LV, Ivanova S, Zhang M, Yang H, Botchkina GI, Watkins LR, Wang H, Abumrad N, Eaton JW, Tracey KJ. Vagus nerve stimulation attenuates the systemic inflammatory response to endotoxin. Nature. 2000 May 25;405(6785):458-62. doi: 10.1038/35013070. PMID 10839541
- [Background] Montano N, Porta A, Cogliati C, Costantino G, Tobaldini E, Casali KR, Iellamo F. Heart rate variability explored in the frequency domain: a tool to investigate the link between heart and behavior. Neurosci Biobehav Rev. 2009 Feb;33(2):71-80. doi: 10.1016/j.neubiorev.2008.07.006. Epub 2008 Jul 30. PMID 18706440
- [Background] Porta A, Gnecchi-Ruscone T, Tobaldini E, Guzzetti S, Furlan R, Montano N. Progressive decrease of heart period variability entropy-based complexity during graded head-up tilt. J Appl Physiol (1985). 2007 Oct;103(4):1143-9. doi: 10.1152/japplphysiol.00293.2007. Epub 2007 Jun 14. PMID 17569773
- [Background] Porta A, Guzzetti S, Montano N, Furlan R, Pagani M, Malliani A, Cerutti S. Entropy, entropy rate, and pattern classification as tools to typify complexity in short heart period variability series. IEEE Trans Biomed Eng. 2001 Nov;48(11):1282-91. doi: 10.1109/10.959324. PMID 11686627
- [Background] Fang J, Egorova N, Rong P, Liu J, Hong Y, Fan Y, Wang X, Wang H, Yu Y, Ma Y, Xu C, Li S, Zhao J, Luo M, Zhu B, Kong J. Early cortical biomarkers of longitudinal transcutaneous vagus nerve stimulation treatment success in depression. Neuroimage Clin. 2016 Dec 18;14:105-111. doi: 10.1016/j.nicl.2016.12.016. eCollection 2017. PMID 28180068
- [Background] Hein E, Nowak M, Kiess O, Biermann T, Bayerlein K, Kornhuber J, Kraus T. Auricular transcutaneous electrical nerve stimulation in depressed patients: a randomized controlled pilot study. J Neural Transm (Vienna). 2013 May;120(5):821-7. doi: 10.1007/s00702-012-0908-6. Epub 2012 Nov 2. PMID 23117749
- See also: Dalle Grave, R., Sartirana, M., & Calugi, S. La gestione dei casi complessi nei disturbi dell'alimentazione. Verona: Positive Press, 2019 — http://www.dallegrave.it/la-gestione-dei-casi-complessi-nei-disturbi-dellalimentazione/
- See also: Eating Disorders: Recognition and Treatment (NICE Guideline 69). — https://www.nice.org.uk/guidance/ng69
- See also: Montano, A. & Flebus, Giovanni Battista. (2006). Presentation of the Beck Depression Inventory - Second edition (BDI-II): Confirmation of bifactorial structure in a sample of the Italian population. — https://www.researchgate.net/publication/294630138_Presentation_of_the_Beck_Depression_Inventory_-_Second_edition_BDI-II_Confirmation_of_bifactorial_structure_in_a_sample_of_the_Italian_population
- See also: CG Fairburn - 2010. La terapia cognitivo comportamentale dei disturbi dell'alimentazione. Firenze, Eclipsi; 2010. — https://books.google.it/books?id=pnJ-OPvhOtoC&lpg=PA1&ots=2U2IeUpAi1&dq=CG%20Fairburn%20-%202010.%20La%20terapia%20cognitivo%20comportamentale%20dei%20disturbi%20dell%E2%80%99alimentazione.%20Firenze%2C%20Eclipsi%3B%202010.&lr&hl=it&pg=PA1#v=onepage&q=CG%20Fairburn%20-%202010.%20La%20terapia%20cognitivo%20comportamentale%20dei%20disturbi%20dell%E2%80%99alimentazione.%20Firenze,%20Eclipsi;%202010.&f=false